CLINICAL TRIAL: NCT02600572
Title: Changes in Attention Level Due to Isometric Exercises and Level Three Progression Eccentric Movements
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics reason at the data collection site
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CI-IRB-20151104003
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Therapy, Exercise
Keywords: balance, postural; postural equilibrium; mental speed; isometric exercise; eccentric exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isometric exercise (Experimental): Subjects performing the isometric exercises intervention
  Interventions: Other: Isometric exercises
- Eccentric exercise (Experimental): Subjects performing the eccentric exercises intervention
  Interventions: Other: Eccentric exercises

INTERVENTIONS:
Other: Isometric exercises — Subjects will perform one session of isometric exercises at the end of Day 1
  Arms: Isometric exercise
Other: Eccentric exercises — Subjects will perform one session of eccentric exercises at the end of Day 2
  Arms: Eccentric exercise

SUMMARY:
Determine the changes in attention level due to isometric exercises and level three progression eccentric movements. The attention level will be measured using a mental speed test (how quickly a subject can process information and make decisions based upon that information). Another outcome measure will be the ability of the subject to maintain balance

DETAILED DESCRIPTION:
On Day 1, subjects will complete the mental speed test and will undergo CDP testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface (a 4" tall foam cushion of known mechanical properties) in a comfortable posture, feet shoulder width, with eyes open or closed, head straight and arms to the side and free to move, gazing forward, and breathing normally. These will constitute the baseline information. Subjects will be divided into two groups: a isometric group (performing the isometric exercises) and an eccentric group (performing the eccentric exercises). At the end of Day 1, the isometric group will perform the isometric exercises while the eccentric group will act as control (no exercise). On Day 2, subjects will complete the mental speed test and will undergo the CDP testing a second time. These will constitute the first follow-up information. At the end of Day 2, the eccentric group will perform the eccentric exercises while the isometric group will act as control (no exercise). Throughout Day 3, subjects will complete the mental speed test and undergo the CDP testing a third time. This will constitute the second and last follow-up information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Any pathology preventing the subject to safely perform the isometric exercises (the clinician enrolling the subjects will make the decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in Stability Score | Baseline, Day 2 and Day 3
  The Stability Score is calculated as percentage ratio of the actual sway and the theoretical limit of stability.
  Changes in Stability Score will be assessed between baseline (Day 1), and Day 2 and Day 3. It will be used to investigate if and which exercises affect it and how much.

SECONDARY OUTCOMES:
Changes in Mental Speed | Baseline, Day 2 and Day 3
  The subject will be presented a series of word/image pairs and/or simple mathematical equations or number sequences. If a pair matches, the subject has to click the "Correct" button, if the pair does not match, the "Incorrect" button . However, if the word "Opposite" appears at the top of the screen, the answer needs to be reversed. The subject has up to 5 minutes to complete the task. The Accuracy of the answers expressed as percentage will be used as measure of mental speed. Changes in Accuracy will be assessed between baseline (Day 1), and Day 2 and Day 3. It will be used to investigate if and which exercises affect it and how much.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies, Cape Canaveral, Florida, United States